CLINICAL TRIAL: NCT02482103
Title: Safety, Success Rate and Long Term Consequences of Renal Denervation in Patients With Therapy Resistant Hypertension. The Dutch National Renal Denervation Registry
Brief Title: The Dutch National Renal Denervation Registry
Acronym: NL_RDN_REG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Principal Investigator, Michiel L. Bots, Professor of Epidemiology of Cardiovascular Disease, UMC Utrecht
Other Study IDs: NL-RDN_REG
Record Dates: First submitted 2015-06-11; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: Therapy resistant hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with renal denervation: Patients treated with RD in the Netherlands. The decision to perform RD was made by the treating physician in the participating hospitals.
  Interventions: Procedure: Renal denervation

INTERVENTIONS:
Procedure: Renal denervation — Catheter based renal nerve ablation

SUMMARY:
This study is a national registry of patients treated with renal denervation (RD) in the Netherlands.

The aim of the study is to collect data on safety of the procedure, predictors of the blood pressure lowering effect, sustainability of the effect and to assess the cardiovascular event rate in patients treated with renal denervation.

This is a prospective observational study.

DETAILED DESCRIPTION:
Hypertension is common and one of the major risk factors for cardiovascular disease. Therefore, it is a major societal and economic health problem. A substantial proportion (20-40%) of the treated hypertensive patients has sub-optimal blood pressure control despite the use of multiple drugs. All these patients have an increased cardio-vascular risk. Furthermore, the use of multiple drugs diminishes compliance to treatment, and increases the risk of side effects. This underscores the need for new approaches for hypertension management. Elevated (renal) sympathetic nerve activity contributes importantly to the development of hypertension and subsequent vascular risk. Deliberate disruption of sympathetic nerve activity (sympatholytic therapy) leads to improvement of vascular outcome through blood pressure dependent and blood pressure independent effects. Recently, a promising novel sympatholytic approach has been introduced, i.e. catheter-based renal denervation in a small clinical trial with resistant hypertensive patients. Many clinical centres have now started to perform this procedure or are in the process to start up.

The Dutch Minister of Health has decided to allow renal denervation in patients with so called resistant hypertension, and "conditional reimbursement" is available starting Jan 1st 2013 for a maximum of 4 years. The Netherlands Organisation for Health Research and Development (ZonMw) has provided us with a grant to perform a randomized trial (SYMPATHY) to evaluate the effect on blood pressure at 6 months after intervention. Maximum follow-up in this trial will be 2 years. Important limitations of this study are, firstly that that follow-up is limited to 2 years after renal denervation. Secondly, not all patients that undergo renal denervation, will participate in the abovementioned trial. The Dutch National Renal Denervation Registry will complement the information from the trial in several aspects. These deal with safety, non-responders, and sustainability.

Objectives of the national database are to collect data that will deliver information on:

Safety:

1. What are the short and long term procedural related complications?

   Responders
2. What are the predictors for the effect on blood pressure, in particular patient related factors and procedural related factors?
3. Are there differences between the various renal denervation devices?

   Sustainability
4. What is the effect on blood pressure after (3), 6, (9), 12, (18), 24, (30), 36, and 60 months and thereafter in patients who are considered eligible based on the judgement of the treating physician?
5. What is the effect on kidney function after (3), 6, (9), 12, (18), 24, (30), 36, and 60 months and thereafter in patients who are considered eligible based on the judgement of the treating physician?
6. What are the cardiovascular events rates in this population, in strata of achieved blood pressure level, and potentially compared with other populations.

Methods:

With this database a nationwide cohort is build comprising patients treated with renal denervation over the years, with uniform baseline data collection and uniform follow-up measurements in terms of safety measurements, blood pressure measurements, hospitalisations, cardiovascular outcomes and all-cause mortality. The data collection will occur through a web-based data entry application. All centers in the Netherlands that perform renal denervation will be asked to participate. All patients who underwent renal denervation should be included, irrespective of the reason and device used.

To address the outstanding research questions specific statistical analyses plans will be applied.

Conclusion:

Our expected results are:

1. to be able to identify patients characteristics, which are associated with a high probability of a favourable blood pressure response to renal denervation,
2. to provide short-and long-term (24 -60 months) side effects of renal denervation

Perspective:

These results, collected in routine clinical practice in a large number of clinics in the Netherlands, will have a major impact on the treatment of 'resistant hypertension'. The safety and efficacy data will pave the way for formal cost-effectiveness analyses. The data have the potential to be of high relevance to decision and policy makers in the government and health insurances. When deemed cost-effective and safe, this approach will be widely used in the treatment of 'resistant hypertension' and will revolutionise the treatment of these patients. Furthermore, it will open ways for evaluation of other groups of patients characterized by a high sympathetic tone; in particular patients with less severe hypertension, heart failure and chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* treated with renal denervation. The decision to perform the procedure was made by the treating physician in the participating hospitals

Exclusion Criteria:

* below age of 18 years

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with (or evaluated and refused for) renal denervation in Dutch hospitals. Indications for RD (by Dutch consensus) are therapy resistant hypertension defined as a blood pressure above treatment goal despite use of 3 or more antihypertensive agents preferably including a diuretic or intolerance for (additional) antihypertensives. Secondary hypertension is excluded beforehand.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-04; Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure | 6 months
  Change in blood pressure at 6 months

SECONDARY OUTCOMES:
safety aspects (change in renal function) | 5 years
  change in renal function
safety aspects: long term kidney function | 5 years
  change in renal function
longterm consequences: CVD events | 5 years
  cardiovascular event rates
safety aspects: procedures complication | 1 year
  procedural complications
longterm consequences: kidney function | 5 years
  change in kidney function
longterm consequences: mortality | 5 years
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michiel L. Bots, MD, PhD, Principal Investigator — Julius Center for Health Sciences and Primary Care
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Vink EE, Bots ML, Blankestijn PJ. Renal denervation as therapy for hypertension: potentials and unanswered questions. Eur J Prev Cardiol. 2013 Dec;20(6):980-91. doi: 10.1177/2047487312473019. Epub 2012 Dec 19. PMID 23610453
- [Result] Verloop WL, Vink EE, Spiering W, Blankestijn PJ, Doevendans PA, Bots ML, Vonken EJ, Voskuil M, Leiner T. Effects of renal denervation on end organ damage in hypertensive patients. Eur J Prev Cardiol. 2015 May;22(5):558-67. doi: 10.1177/2047487314556003. Epub 2014 Oct 17. PMID 25326543
- [Result] Vink EE, Verloop WL, Bost RB, Voskuil M, Spiering W, Vonken EJ, Bots ML, Blankestijn PJ. The blood pressure-lowering effect of renal denervation is inversely related to kidney function. J Hypertens. 2014 Oct;32(10):2045-53; discussion 2053. doi: 10.1097/HJH.0000000000000282. PMID 25023158
- [Result] Verloop WL, Vink EE, Spiering W, Blankestijn PJ, Doevendans PA, Bots ML, Vonken EJ, Voskuil M. Renal denervation in multiple renal arteries. Eur J Clin Invest. 2014 Aug;44(8):728-35. doi: 10.1111/eci.12289. PMID 24931208
- [Result] Verloop WL, Vink EE, Voskuil M, Vonken EJ, Rookmaaker MB, Bots ML, Doevendans PA, Blankestijn PJ, Spiering W. Eligibility for percutaneous renal denervation: the importance of a systematic screening. J Hypertens. 2013 Aug;31(8):1662-8. doi: 10.1097/HJH.0b013e328362152e. PMID 23743806
- [Result] Persu A, Jin Y, Baelen M, Vink E, Verloop WL, Schmidt B, Blicher MK, Severino F, Wuerzner G, Taylor A, Pechere-Bertschi A, Jokhaji F, Fadl Elmula FE, Rosa J, Czarnecka D, Ehret G, Kahan T, Renkin J, Widimsky J Jr, Jacobs L, Spiering W, Burnier M, Mark PB, Menne J, Olsen MH, Blankestijn PJ, Kjeldsen S, Bots ML, Staessen JA; European Network Coordinating research on REnal Denervation Consortium. Eligibility for renal denervation: experience at 11 European expert centers. Hypertension. 2014 Jun;63(6):1319-25. doi: 10.1161/HYPERTENSIONAHA.114.03194. Epub 2014 Mar 24. PMID 24664290